CLINICAL TRIAL: NCT05739708
Title: Psychological Characteristics of Patients With Severe Asthma
Acronym: CATAPLASTHMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/727
Record Dates: First submitted 2023-02-02; First posted 2023-02-22 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Asthma; Attachment; Coping Skills; Personality Trait
MeSH Terms: conditions — Asthma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthma patients (Other)
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The time to complete the different questionnaires is estimated to be 60 minutes.
  Other Names: Asthma Coping List (French version); Big Five Inventory (French version); Relationship Scales Questionnaire (French version); Hospital Anxiety and Depression Scale (French version); Asthma Quality of Life Questionnaire (French version); Working Alliance Inventory-Short Form Revised (French version); Asthma Control Test (French version); Morisky Medication Adherence Scale (French version)

SUMMARY:
Like any chronic disease, asthma exposes individuals to stressful and threatening situations that require ongoing cognitive, emotional, behavioral and social adaptation. Approximately 5-10% of patients with asthma have a treatment-resistant disease, with frequent emergency room visits and hospitalizations. These patients are responsible for the majority of the overall asthma-related disease burden and also represent more than half of the total direct costs of asthma management. The scientific literature shows that personality traits, attachment type and psychological disorders will significantly influence disease coping strategies, disease experience, quality of life, adherence and therapeutic alliance. Although some data exist in asthma, there are currently no studies that have evaluated the overall psychological profile of asthma patients, and we have no data specifically on the population of severe asthmatics, who are the most difficult to manage. A better understanding of the overall psychological dimension of asthma patients will make it possible to offer therapeutic education programs that are more targeted according to the psychosocial skills of the patient and finally improve the overall management of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years and followed in the Respiratory Department of the Besançon University Hospital for an asthmatic disease diagnosed for more than 12 months. Will be considered as severe patients, asthma patients with uncontrolled asthma despite high therapeutic pressure (GINA levels 4 and 5) and patients requiring to be controlled high doses of inhaled corticosteroids and long-acting beta-2-agonists (or anti-leukotriene/theophylline) in the past year or systemic corticosteroid therapy (>50% in the previous year) (ATS-ERS 2014 criteria).
* Patient able to understand the objectives of the research
* Patient who has signed a research consent form
* Patient affiliated to a French social security system or beneficiary of such a system

Exclusion Criteria:

* Patient with reading and comprehension difficulties that prevent them from completing the questionnaires
* Motor disability that prevents the patient from completing the questionnaires
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and/or poor cooperation anticipated by the the investigator
* Subject without health insurance
* Subject under court protection, guardianship, conservatorship, or protective supervision. protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Description of the psychological profile of severe asthma patients | 1 day
  Score on questionnaires assessing coping strategies (ACL-F)
Description of the psychological profile of severe asthma patients | 1 day
  Score on questionnaire personality traits (BFI-Fr)
Description of the psychological profile of severe asthma patients | 1 day
  Score on questionnaire attachment types (RSQ)
Description of the psychological profile of severe asthma patients | 1 day
  Score on questionnaire anxiety and depression (HADS)
Description of the psychological profile of severe asthma patients | 1 day
  Score on questionnaire quality of life (AQLQ)
Description of the psychological profile of severe asthma patients | 1 day
  Score on questionnaire patient-physician therapeutic alliance (WAI-SR)
Description of the psychological profile of severe asthma patients | 1 day
  Score on questionnaire 0Asthma Control Test (ACT)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon - Service de Pneumologie, Besançon, Doubs, France